CLINICAL TRIAL: NCT02165358
Title: Muscle MRI Study of Patients With Becker Muscular Dystrophy and Limb-girdle Muscular Dystrophy Type 2I
Brief Title: Muscle MRI in Becker Muscular Dystrophy and in Limb-girdle Muscular Dystrophy Type 2I
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Nicoline Løkken, Bsc, Rigshospitalet, Denmark
Other Study IDs: H-2-2014-035 (MRI BMD/LGMD2I)
Record Dates: First submitted 2014-06-11; First posted 2014-06-17 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Becker Muscular Dystrophy; Limb-Girdle Muscular Dystrophy Type 2I
Keywords: BMD; LGMD2I; Calf enlargement; Muscular dystrophy; MRI
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophy, Limb-Girdle, Type 2I; Muscular Dystrophies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Patients verified with either becker muscular dystrophy or limb-girdle muscular dystrophy type 2I
- Controls: Healthy controls matched for age and gender.

SUMMARY:
The purpose of this study is to investigate the paradoxical muscle enlargement in the calves and tongue seen in patients affected by Becker muscular dystrophy and Limb-girdle muscular dystrophy type 2I.

The enlarged calves' muscle quality will be assessed primarily on the basis of the muscle structure on MRI and based on a calculation of muscle strength per cross-sectional area.The findings will be compared with results from non-affected controls.

Additionally we want to describe the tongue muscle appearance on T1-weighted MRI.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the paradoxical muscle enlargement seen in patients affected by Becker muscular dystrophy and Limb-girdle muscular dystrophy type 2I.

Becker and limb-girdle muscular dystrophies are both hereditary muscular disorders. Both diseases appear clinically with shrinkage and muscle weakness of the muscles around the shoulder girdle and pelvis, while muscle hypertrophy of the calves and tongue is seen.

The quality of the enlarged calves has to the investigators knowledge not previously been described, and their hypothesis is that the normal correlation between muscle strength and muscle cross-section is absent in the calf muscles. Thus the investigators hypothesis suggests that there is no actual hypertrophy of the calf muscles, but rather a pseudohypertrofy with reduced force per cross-sectional area. With a picture of increased fat infiltration and disorganized muscle fibers.

The enlarged calves' muscle quality will be assessed primarily on the basis of the muscle structure on MRI (assessed on both T1 imaging, 3-point Dixon scans, and diffusion tension imaging), and based on a calculation of muscle strength per cross-sectional area. Isokinetic muscle dynamometry (Biodex-4) will be used to measure muscle strength. The findings will be compared with results from non-affected controls.

Additionally the investigators want to describe the tongue muscle appearance on T1-weighted MRI.

ELIGIBILITY:
Inclusion Criteria:

* Danish patients genetically verified with either becker muscular dystrophy or limb-girdle muscular dystrophy type 2I
* calves enlargement

Exclusion Criteria:

* Patients who have metal implants in the body, for instance surgical clips, cochlear implants, pacemaker etc.
* pregnant or breast-feeding patients
* patients who are claustrophobic
* atrophic calves

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Danish patients genetically verified with either becker muscular dystrophy or limb-girdle muscular dystrophy type 2I
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Calves muscle quality | 1 day
  the investigators will describe muscle quality by:
  1. MRI scans of the calves comprising of a T1-weighted MRI scan, a 3-point Dixon scan to measure the fraction of fat in the muscle, a short TI inversion recovery (STIR) scan, and a diffusion tensor imaging (DTI) scan to see the muscle fiber organization.
     The MRI scans will further be used to measure the fat free muscle cross-sectional area of the muscle groups responsible for plantar flexion and dorsi flexion respectively.
  2. Biodex muscle strength measurements: Isokinetic muscle dynamometry measurements on plantar flexion and dorsal flexion over the ankle.
  3. Calculating of muscle strength per muscle cross-sectional area

SECONDARY OUTCOMES:
MRI T1 scan of the tongue | 1 day
  MRI T1 scan of the tongue to investigate muscle volume

CONTACTS AND LOCATIONS:
Overall Officials: Nicoline Løkken, Bsc, Principal Investigator — Neuromuscular Research Unit, Rigshospitalet, Copenhagen
Locations (1):
- Neuromuscular Research Unit, Rigshospitalet, Copenhagen, Denmark